CLINICAL TRIAL: NCT04188392
Title: Pilot Feasibility Study of Pimavanserin for Insomnia in Veterans With Posttraumatic Stress Disorder
Brief Title: Pimavanserin for Insomnia In Veterans With Posttraumatic Stress Disorder
Acronym: PIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Melissa Jones, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-45799
Record Dates: First submitted 2019-12-04; First posted 2019-12-05 (Actual); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Post-traumatic Stress Disorder; Insomnia
Keywords: Post-traumatic Stress Disorder; Insomnia
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders | interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- open-label treatment (Experimental): pimavanserin 34mg at bedtime for 6 weeks
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — pimavanserin tablet
  Other Names: Nuplazid

SUMMARY:
This preliminary, open-label study assesses the feasibility of 34mg at bedtime for 6 weeks in Veterans with Posttraumatic Stress Disorder and insomnia.

DETAILED DESCRIPTION:
More treatments are needed to target insomnia in Veterans with Posttraumatic Stress Disorder. There is evidence to suggest that pimavanserin, a medication approved by the Food and Drug Administration for the treatment of psychosis in Parkinson's disease, may improve deep sleep and insomnia. This study preliminary assesses the feasibility of pimavanserin 34mg at bedtime for 6 weeks for the treatment of chronic insomnia in Veterans with Posttraumatic Stress Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for current Posttraumatic Stress Disorder (PTSD), as per a total score of ≥33 on the PTSD Checklist (PCL-5) and Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-5) criteria for PTSD.
* Meets DSM-5 standards of chronic insomnia disorder, as follows: a. Complains of dissatisfaction with nighttime sleep in the form of difficulty falling asleep (subjective sleep onset latency ≥30 minutes), difficulty staying asleep (subjective time awake after sleep onset ≥30 minutes), and/or awakening earlier in the morning (≥30 minutes before scheduled wake time and before a total sleep time of 6.5 hours) than desired. b. Insomnia frequency of ≥3 times per week c. The duration of the insomnia complaint is ≥3 months d. Associated with complaint of daytime impairment.
* Insomnia Severity Index total score ≥15 (moderate insomnia).
* Willing to not start a concurrent behavioral or other treatment program for insomnia, PTSD, or other psychiatric disorders during the participation in the study.
* Women of child-bearing potential who are sexually active agree to use two methods of contraception for the duration of the study and extending to 30 days after the last dose of study drug.

Exclusion Criteria:

* Current or a history of a primary psychotic disorder (i.e., schizophrenia, schizoaffective or bipolar disorder)
* Active suicidal or homicidal ideation requiring crisis intervention
* Current moderate or severe alcohol or marijuana use disorder, or other illicit use disorder of any severity
* A history of moderate or severe traumatic brain injury or other neurological illness (i.e., stroke, epilepsy, multiple sclerosis);
* Caffeine use that is deemed excessive and is contributing to the insomnia per the opinion of the investigators (i.e. caffeinated beverages consumed after 18:00 3 times/week or more and/or that correlates with the timing of the insomnia complaints).
* Tobacco use before bedtime that is contributing to the insomnia per the opinion of the investigators or that would interfere with completing an overnight polysomnogram.
* Previous diagnosis of periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, narcolepsy, Rapid Eye Movement Behavior Disorder, or other sleep disorders (except obstructive sleep apnea) that may confound, per the opinion of the investigators, the assessment of insomnia.
* Previous diagnosis of moderate to severe obstructive sleep apnea (defined as an AHI equal to or greater than 15)
* Participants deemed to be at high risk of moderate to severe obstructive sleep apnea per the Snoring, Tiredness, Observed apnea, high blood Pressure, Body mass index, Age, Neck circumference, and male Gender questionnaire (STOP-BANG). Subjects with a STOP-BANG score of 5 or greater, or STOP score of 2 or greater plus body mass index greater than 35 kg/m2 or male or neck circumference greater than 40 cm, are considered to be high-risk. These participants can re-enter the study following adherence to therapy for 1-month and if inclusion and exclusion criteria are still met.
* Participants identified as having moderate to severe obstructive sleep apnea during the screening polysomnogram. These participants will be referred to clinical treatment
* Periodic limb movement arousal index 15 or greater or other sleep disorders captured during the screening polysomnogram that may confound, per the opinion of the investigators, the assessment and treatment of insomnia
* A prolonged QT interval, corrected for heart rate (QTc), at the screening electrocardiogram. A prolonged QTc is defined as 470 milliseconds for males and 480 milliseconds for females.
* Engagement in an evidence-based psychotherapy for 1-week prior to enrollment that in the opinion of the investigators, may confound the assessment of insomnia
* Current evidence of clinically significant cardiac, respiratory, gastrointestinal, renal, neurological, hepatic, and/or chronic pain that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Females who are breastfeeding or pregnant at screening
* Females of childbearing potential who are not practicing acceptable pregnancy prevention methods (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal or have been sterilized surgically).
* Current use of a prohibited medications: Hypnotic or sedating medications taken at bedtime for insomnia; antipsychotics and antidepressants with known 5HT2A antagonist activity; medications that increase or decrease the metabolism of pimavanserin; medications that increase the risk of QTc prolongation
* Patients with conditions known to increase the risk of torsades de pointes and/or sudden death, such as symptomatic bradycardia and other cardiac arrhythmias, uncorrected hypokalemia or hypomagnesemia, and congenital prolongation of the QT interval.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa B Jones, MD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Patient health information will not be transmitted to collaborators.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from clinics and clinician referrals at the Michael E. DeBakey VA Medical Center
Pre-assignment Details: Pre-assignment exclusions (n=5): non-adherent to CPAP (n=2), bradycardia and hepatic dysfunction (n=1), psychosis (n=1), lost to follow up (n=1)
Period: Overall Study
Arm/Group | Open-label Treatment
Started | 6
Sleep Studies 1 and 2 | 6
Mid-point Visit (Treatment Week-3) | 6
Sleep Study 3 | 5 (1 subject could not complete sleep study 3 due to hospital-wide shut-downs during the COVID pandemic.)
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects enrolled into open-label treatment
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.33 (6.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Current depressive disorder [Count of Participants; unit: Participants] — Current depressive disorder per the Structured Clinical Interview for the DSM-5
  Participants | 4

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rates
Description: The rate of enrollment per month; goal of 6 subjects total
Time Frame: Total duration of recruitment time (5.8 months)
Population: Subjects enrolled into open label treatment
Measure: Mean (95% Confidence Interval); unit: participants enrolled per month
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
participants enrolled per month | 1.03 [0.38 to 2.25]
Statistical Analysis 1: Comparison: Open-label Treatment; Recruitment goal of 6 subjects total; Test type: Other — Rate of subjects enrolled per month of recruitment; based on 6 subjects enrolled over 5.8 months of recruitment; Rate (per month) = 1.03, 95% CI 2-sided [0.38 to 2.25] — Based on 6 subjects enrolled over 5.8 months of recruitment

2. Primary Outcome: Retention Rates
Description: The number of subjects who complete the protocol in its entirety; goal of 75% of subjects enrolled into treatment
Time Frame: 10 weeks (overall study)
Population: Subjects enrolled into open-label treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
Participants | 6
Statistical Analysis 1: Comparison: Open-label Treatment; Binary outcome (completed protocol yes vs. no); goal of 75% of subjects completing protocol; Test type: Other — Total participants = 6; completed protocol: yes = 6, no = 0; Point estimate = 1, 95% CI 2-sided [0.54 to 1] — Point estimate = 100% (95% C.I. 54%,100%); Point estimate of completion rate and 95% confidence interval

3. Secondary Outcome: Mean Change in Duration of Stage N3 Sleep Pre- and Post-treatment
Description: The mean difference in duration of stage N3 sleep from baseline polysomnogram to week-6 polysomnogram ([Time in N3 post-treatment] - [Time in N3 at baseline polysomnogram])
Time Frame: 6 weeks (time between baseline and closeout polysomnogram)
Population: Subjects enrolled in open-label treatment and completed baseline and post-treatment polysomnogram (1 subject could not complete post-treatment polysomnogram due to pandemic).
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 5
minutes | 21.7 (39.57)
Statistical Analysis 1: Comparison: Open-label Treatment; alternative hypothesis: true difference in means is not equal to 0; Test type: Other — paired t-test; p = 0.2873, t-test, 2 sided — A priori significance threshold of p<0.05; t=1.2263, df=4; Mean of the differences = 21.7, 95% CI 2-sided [-27.4 to 70.8]

4. Secondary Outcome: Discontinuation Rates Due to Adverse Effects
Description: The number of subjects who discontinue the protocol due to adverse effects (from either protocol or medication)
Time Frame: 10 weeks (overall study duration)
Population: Number of subjects enrolled into open-label treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
Participants | 0
Statistical Analysis 1: Comparison: Open-label Treatment; Binary outcome: Discontinued due to adverse effects yes vs. no; Test type: Other — Total participants = 6; discontinued due to adverse effects: yes = 0, no =6; Point estimate, 95% confidence interval = 0, 95% CI 2-sided [0 to 0.46] — Discontinuation rates due to adverse effects: Point estimate 0% (95% C.I. 0%, 45.9%)

5. Secondary Outcome: Completion Rates of Key Outcome Measures
Description: The percentage of participants who complete subject and objective measures of insomnia, including sleep diaries, actigraphy, and attended polysomnography
Time Frame: 10 weeks (overall study duration)
Population: Subjects enrolled into open-label treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
Participants
  Completed sleep study 1 | 6
  Completed sleep study 2 | 6
  Completed sleep study 3 | 5
  At least 4 days of actigraphy pre-treatment | 6
  At least 4 days of actigraphy post-treatment | 6
  At least 4 days of sleep diary pre-treatment | 6
  At least 4 days of sleep diary post-treatment | 6
Statistical Analysis 1: Comparison: Open-label Treatment; Binary outcome: Completed sleep study 1 yes vs. no; Test type: Other — Total participants = 6; completed sleep study 1: yes = 6, no=0; point estimate = 1, 95% CI 2-sided [0.54 to 1] — Point estimate of completion rate for sleep study 1 = 100% (95% C.I. 54%, 100%)
Statistical Analysis 2: Comparison: Open-label Treatment; Binary outcome: completed sleep study 2 yes vs. no; Test type: Other — Total participants = 6; completed sleep study 2: yes = 6, no=0; point estimate = 1, 95% CI 2-sided [0.54 to 1] — Point estimate of completion rate for sleep study 2 = 100% (95% C.I. 54%, 100%)
Statistical Analysis 3: Comparison: Open-label Treatment; Binary outcome: completed sleep study 3 yes vs. no; Test type: Other — Total participants = 6; completed sleep study 3: yes = 5, no=1; point estimate = 0.83, 95% CI 2-sided [0.36 to 0.996] — Point estimate of completion rate for sleep study 3 = 83.3% (95% C.I. 36%, 99.6%)
Statistical Analysis 4: Comparison: Open-label Treatment; Binary outcome: at least 4 days of actigraphy data pre-treatment yes vs. no; Test type: Other — Total participants = 6; at least 4 days of actigraphy data: yes = 6, no=0; point estimate = 1, 95% CI 2-sided [0.54 to 1] — Point estimate of completion rate for at least 4 days of actigraphy pre-treatment = 100% (95% C.I. 54%, 100%)
Statistical Analysis 5: Comparison: Open-label Treatment; Binary outcome: at least 4 days of actigraphy post-treatment yes vs. no; Test type: Other — Total participants = 6; at least 4 days of actigraphy post-treatment: yes = 6, no =0; point estimate = 1, 95% CI 2-sided [0.54 to 1] — Point estimate of at least 4 days of actigraphy post-treatment = 100% (95% C.I. 54%, 100%)
Statistical Analysis 6: Comparison: Open-label Treatment; Binary outcome: at least 4 days of sleep diary pre-treatment yes vs. no; Test type: Other — Total participants = 6; at least 4 days of sleep diary pre-treatment: yes = 6, no = 0; point estimate = 1, 95% CI 2-sided [0.54 to 1] — Point estimate of at least 4 days of sleep diary pre-treatment = 100% (95% C.I. 54%, 100%)
Statistical Analysis 7: Comparison: Open-label Treatment; Binary outcome: at least 4 days of sleep diary post-treatment yes vs. no; Test type: Other — Total participants = 6; at least 4 days of sleep diary post-treatment: yes = 6, no = 0; point estimate = 1, 95% CI 2-sided [0.54 to 1] — Point estimate of at least 4 days of sleep diary post-treatment = 100% (95% C.I. 54%, 100%)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Assessed with staff-administered questionnaire at all in-person and telephone visits following enrollment
Arm/Group | Open-label Treatment
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Treatment (N=6)
skin irritation (Skin and subcutaneous tissue disorders) | 3 — From actigraphy watch
skin irritation (Skin and subcutaneous tissue disorders) | 1 — From sleep study tubing
sleepiness (General disorders) | 2 — Mild sleepiness that resolved after first dose
dry mouth (General disorders) | 1
headache (Nervous system disorders) | 1 — Similar in frequency and intensity to historical headaches and deemed by investigators to be unrelated to medication
arthralgia (Musculoskeletal and connective tissue disorders) | 1 — Deemed by investigators to be unrelated to medication
diarrhea (Gastrointestinal disorders) | 1 — Associated with brief gastrointestinal illness deemed by investigators to be unrelated to medication
weight gain (General disorders) | 1 — Deemed by investigators to be unrelated to medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT04188392/Prot_SAP_ICF_000.pdf